CLINICAL TRIAL: NCT07378683
Title: A Prospective, Single-Center Clinical Validation Study: Machine Learning Model-Based Risk Stratification Intervention for Reducing Surgical Site Infection After Central Nervous System Tumor Surgery
Brief Title: A Clinical Prediction Model for Surgical Site Infection After Central Nervous System Tumor Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ming Yang (Other)
Responsible Party: Sponsor-Investigator, Ming Yang, Clinical Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NCC2025-CNS-SSI; 2024-I2M-3-014 (Other: CAMS Innovation Fund for Medical Sciences)
Record Dates: First submitted 2026-01-22; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Surgical Site Infection (SSI); Central Nervous System Tumor
Keywords: surgical site infection; central nervous system tumor; machine learning; explainable artificial intelligence; SHAP; clinical decision support system
MeSH Terms: conditions — Surgical Wound Infection; Central Nervous System Neoplasms

STUDY DESIGN:
Intervention Model Description: A prospective, single-center clinical validation study aimed at evaluating the effectiveness of a machine learning (LightGBM) model-based risk stratification intervention strategy in reducing the incidence of surgical site infection (SSI) in patients after central nervous system tumor surgery.
  The study plans to enroll 500 patients undergoing elective surgery. SSI risk will be calculated within 72 hours postoperatively using the model, which is based on 8 clinical features. The high-risk group (predicted probability ≥50%) will receive individualized enhanced interventions (e.g., antibiotic escalation, nutritional support), while the low-risk group (predicted probability <50%) will receive standard care. The primary endpoint is the incidence of SSI within 90 days postoperatively (NHSN criteria), and secondary endpoints include model performance, hospital stay length, medical costs, etc.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Risk: ML-Based Intervention (Experimental): This is the High-Risk Intervention Group. Patients identified as high-risk for SSI (predicted probability ≥ 50%) by the LightGBM model within 72 hours post-surgery receive an enhanced, individualized intervention package, which may include an escalated antibiotic regimen, intensified nutritional support, and closer monitoring.
  Interventions: Other: ML-Based Enhanced Intervention Package for SSI Prevention
- Low-Risk: Standard Care (Active Comparator): This is the Low-Risk Routine Care Group. Patients identified as low-risk for SSI (predicted probability < 50%) by the same model receive the current standard postoperative care of the hospital, following established clinical pathways without the enhanced intervention package. This arm serves as the control.
  Interventions: Other: Standard Postoperative Care

INTERVENTIONS:
Other: ML-Based Enhanced Intervention Package for SSI Prevention — This is a comprehensive, individualized intervention package administered to patients identified as high-risk for surgical site infection (SSI) by a machine learning (LightGBM) model. The package is activated postoperatively and may include, but is not limited to: 1) **Escalated/optimized antibiotic prophylaxis regimen**; 2) **Intensified nutritional support protocols**; 3) **Enhanced monitoring** of vital signs and wound status. The specific components are tailored based on the patient's risk profile and clinical context. The intervention aims to validate the effectiveness of a model-driven strategy in reducing SSI incidence.
  Arms: High-Risk: ML-Based Intervention
Other: Standard Postoperative Care — This intervention represents the current standard of care provided to patients after elective central nervous system tumor surgery at this institution. It includes routine antibiotic prophylaxis, standard wound care, basic vital signs monitoring, and follow-up according to established clinical pathways. Patients in this group do not receive the enhanced, study-specific intervention package and serve as the control population for comparison.
  Arms: Low-Risk: Standard Care

SUMMARY:
1. Study Background For patients undergoing brain or spinal tumor surgery, postoperative surgical wound infection (known as "surgical site infection," SSI) is a recognized risk. Once an infection occurs, it may complicate and prolong the recovery process. Currently, doctors primarily rely on clinical experience to judge which patients are at higher risk of infection. Our research team has previously developed an intelligent prediction model (a machine learning tool) that can very accurately identify which patients are at higher risk of postoperative infection. This study aims to validate whether implementing enhanced preventive measures for high-risk patients in advance, based on the model's predictions, can effectively reduce the occurrence of infection.
2. Study Purpose The primary purpose of this study is to validate whether an individualized intervention strategy based on an intelligent prediction model can effectively reduce the incidence of surgical site infection in patients after central nervous system tumor surgery. Simultaneously, we will also evaluate the safety of this strategy, its impact on patient hospital stay length and medical costs, as well as its feasibility in practical clinical application.
3. Study Design Type: This is a prospective, single-center clinical validation study. "Prospective" means the research plan is established first, followed by patient recruitment and data collection according to the plan; "single-center" indicates the study is conducted solely at the Chinese Academy of Medical Sciences Cancer Hospital.

   Process: For all patients who consent to participate in this study, within 72 hours after surgery, the research system will automatically calculate their infection risk based on 8 key clinical indicators (such as blood test results, medical history, etc.).

   High-Risk Group (model-predicted infection probability ≥50%): Will receive a set of enhanced, individualized infection prevention measures (e.g., adjusted antibiotic regimen, enhanced nutritional support, closer monitoring).

   Low-Risk Group (model-predicted infection probability <50%): Will receive the current standard, high-quality postoperative care.

   Duration: The study is planned to run from February 2026 to October 2029. Each participating patient will be followed for 3 months (90 days) to observe whether infection occurs.

   Sample Size: It is planned to recruit approximately 500 eligible patients.
4. Primary Evaluation Indicators Primary Indicator: The incidence of surgical site infection within 90 days after surgery. The diagnosis of infection will be made by experts who are unaware of the patient's group assignment, strictly following international standards.

   Secondary Indicators: Include the accuracy of the intelligent prediction model in practical use, patient hospital stay length, other infection-related complications, medical costs, and the adoption rate of the model's recommendations by physicians.
5. Eligibility Criteria (Inclusion Criteria Summary)

   You may be eligible to participate in this study if you meet the following conditions:

   Diagnosed with a brain or spinal tumor and scheduled for elective surgery. Aged 18 years or older. Expected survival exceeds 3 months and able to cooperate with postoperative follow-up.

   Voluntary participation and signing of a written informed consent form. (Note: This study has detailed exclusion criteria. Final confirmation of whether all criteria are met will be determined by your study doctor.)
6. Patients' Rights and Safety Voluntary Participation: Participation in this study is entirely voluntary. You have the right to withdraw from the study at any time, which will not affect the quality of any normal medical services you are entitled to at our hospital or your relationship with it.

   Informed Consent: Before the study begins, your study doctor will explain all study procedures, potential risks, and benefits in detail, and you will sign an "Informed Consent Form." Privacy Protection: All your personally identifiable information will be kept strictly confidential. Codes will replace your name and other identifiable information in research analyses and reports.

   Safety Assurance: This study has been reviewed and approved by the hospital's Ethics Committee. We have established an independent Data Safety Monitoring Board to monitor the study's safety throughout. Clinical trial liability insurance has been purchased for all participants to cover damages related to the trial.
7. Contact Information

If you would like to learn more about this study, please contact us via:

Principal Investigator: Dr. Yang Ming National Cancer Center/National Clinical Research Center for Cancer/Cancer Research Unit: Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a pathologically confirmed primary or metastatic central nervous system (brain or spinal) tumor.
2. Scheduled for elective craniotomy or spinal tumor resection surgery.
3. Age ≥ 18 years.
4. Expected survival > 3 months, and able/willing to comply with postoperative follow-up.
5. Voluntary participation and provision of written informed consent.

Exclusion Criteria:

1. Presence of active systemic or local surgical site infection before surgery.
2. Use of therapeutic antibiotics for any reason within 72 hours prior to surgery.
3. Concurrent severe immunosuppressive conditions, or chronic use of high-dose immunosuppressants.
4. Pregnancy or lactation.
5. Known contraindications or severe allergy to the antibiotics planned for use in the study.
6. Any other condition that, in the investigator's judgment, may affect study participation or outcome assessment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2029-10-30 (Estimated); Study Completion 2029-10-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of surgical site infection within 90 days postoperatively | 90 days post-surgery
  The occurrence of a surgical site infection (SSI) following central nervous system tumor surgery, diagnosed according to the U.S. National Healthcare Safety Network (NHSN) criteria. Diagnosis will be adjudicated by a blinded independent endpoint adjudication committee.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, PUMC, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the results reported in this article (including demographics, clinical characteristics, model input variables, and primary endpoint) will be shared. The study protocol, statistical analysis plan, and informed consent form will also be made available. Data will become available following publication of the primary results in a peer-reviewed journal and will be accessible for at least 5 years. Access will be granted to researchers whose methodologically sound proposals have been approved by a scientific review committee, via a controlled-access data repository or upon request.
Supporting Information: Analytic Code
Time Frame: The de-identified IPD and supporting documents will become available no later than 6 months after the publication of the primary study findings in a peer-reviewed journal. The data will be accessible for a minimum of 5 years thereafter.
Access Criteria: Access to IPD will be granted to qualified researchers for legitimate scientific research purposes. Requestors must submit a methodologically sound research proposal to the study Principal Investigator (PI) for review by a designated scientific committee. Proposals will be evaluated for scientific merit, feasibility, and ethical compliance. Data requestors will be required to sign a data use agreement (DUA) prohibiting re-identification attempts, unauthorized redistribution, and commercial use.